CLINICAL TRIAL: NCT05045612
Title: Antibiotic Therapy in Viral Airway Infections: An Open Labeled Randomized Controlled Pragmatic Trial to Evaluate the Efficacy and Safety of Discontinuing Antibiotic Therapy in Adult Patients With Respiratory Viruses
Brief Title: Antibiotic Therapy in Viral Airway Infections
Acronym: ATHENIAN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Magnus Nakrem Lyngbakken, Postdoctoral fellow, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213847; 2021-004248-11 (EudraCT Number)
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Infectious Disease; Influenza; Respiratory Syncytial Virus (RSV); Respiratory Tract Infections
Keywords: pragmatic trial; antibiotic stewardship; viral respiratory tract infection
MeSH Terms: conditions — Communicable Diseases; Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Two-arm, open label, pragmatic randomized controlled non-inferiority stop trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Stop antibiotic therapy as instituted by admitting physician
  Interventions: Other: Stop antibiotic therapy
- Control (No Intervention): Continue antibiotic therapy at the discretion of the treating physician (no change in ongoing treatment)

INTERVENTIONS:
Other: Stop antibiotic therapy — Stop antibiotic therapy instituted by the admitting physician
  Arms: Intervention

SUMMARY:
Antimicrobial resistance is one of the most urgent health threats of our time, and Norwegian hospitals were required to reduce the use of broad-spectrum antibiotics with 30% by the end of 2020. In the current proposal, the investigators aim to assess the efficacy and safety of early discontinuation of antibiotic therapy in adult patients infected with respiratory viruses.

A general recommendation to treat all instances of community acquired pneumonia (CAP) patients with antibiotics leads to significant antibiotic overtreatment. In 2008, the US Food and Drug Administration approved the first multiplex polymerase chain reaction assay for the detection of multiple respiratory virus nucleic acids simultaneously. The wide availability of such nucleic acid amplification tests (NAAT) for rapid viral detection together with chest radiographs has the potential to define patients who can be managed without antibiotics.

Akershus University Hospital is one of the largest hospitals in Norway, with a catchment area of more than 550,000 people. In 2012 to 2013, the majority of patients admitted to Akershus University Hospital with suspected CAP and a positive viral NAAT were treated with antibiotics, a prescription pattern representing antibiotic overtreatment. The investigators accordingly hypothesize that discontinuation of antibiotic therapy in patients with moderately severe disease and airway sample positive for respiratory viruses is safe and non-inferior to continuation of antibiotic therapy.

DETAILED DESCRIPTION:
In patients with positive airway sample for respiratory viruses, the investigators hypothesize that discontinuation of antibiotic therapy is safe and non-inferior to continuation of antibiotic therapy. More specifically, the investigators hypothesize that the early clinical response assessed at 120 hours after randomization, defined as survival with symptom improvement without receipt of rescue antibacterial therapy, will be similar between patients who discontinue and continue antibiotic therapy. Furthermore, the investigators hypothesize that discontinuation of antibiotic therapy is associated with similar mortality rates, duration of hospital admission and reduced number of defined daily doses of antibiotics.

The primary aim is to assess whether discontinuation of antibiotic therapy in patients with positive airway sample for respiratory viruses is safe and associated with early clinical response assessed at 120 hours after randomization that is comparable to patients who continue antibiotic therapy.

The secondary aims are to assess whether discontinuation of antibiotic therapy in patients with positive airway sample for respiratory viruses is associated comparable (1) mortality rates, (2) duration of hospital admission, (3) defined daily doses of antibiotic therapy.

Specific objectives In patients with positive airway sample for respiratory viruses, assess the impact of discontinuing antibiotic therapy on early clinical response quantified as survival with symptom improvement without receipt of rescue antibacterial therapy. Early clinical response is defined as improvement of one or more levels relative to baseline in two or more symptoms of the investigator's assessment of symptoms of community-acquired bacterial pneumonia and no worsening of one or more levels in other symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized
* Adults 18 year or older
* Moderately severe disease (CRB65 ≤ 2 at time of inclusion)
* Nasopharyngeal swab positive for influenza virus, parainfluenza virus, respiratory syncytial virus (RSV) or human metapneumovirus (hMPV)
* On antibiotic therapy as instituted by the receiving physician from the emergency department
* Signed informed consent must be obtained and documented according to ICH GCP, and national/local regulations.

Exclusion Criteria:

* Requiring ICU admission at screening
* Requiring high-flow oxygen therapy or non-invasive ventilation at screening
* Signs of severe pneumonia (abscesses, massive pleural effusion, a well-defined lobar infiltrate on chest X-ray strongly suggestive of bacterial etiology)
* Not immunocompetent (i.e. on active chemotherapy, corticosteroid therapy equaling ≥ 20 mg prednisolone daily for ≥ 4 weeks, chronic immunosuppression due to solid organ transplant)
* SARS-CoV-2 positive
* Bacteremia
* Urine antigen test positive for legionella
* Any other infection necessitating antibiotic treatment
* Antibiotic use for assumed airway infection within the last 24 hours before admission to hospital
* Time from initiation of antibiotic therapy to screening >48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Early clinical response | 120 hours after randomization
  Survival with symptom improvement without receipt of rescue antibacterial therapy

SECONDARY OUTCOMES:
In-hospital mortality | Untill hospital discharge (commonly 3-5 days)
  Mortality during hospital admission
30-day mortality | 30 days after hospital discharge
  Mortality at 30 days after hospital discharge
Duration of hospital admission | Untill hospital discharge (commonly 3-5 days)
  Duration of hospital admission
Antimicrobial days of therapy | Untill hospital discharge (commonly 3-5 days)
  Number of days on antibiotic therapy
Rescue antibiotic therapy during hospital admission | Untill hospital discharge (commonly 3-5 days)
  Rescue antibiotic therapy given to patients randomized to intervention
New antibiotic therapy for presumed airway infection | 30 days after hospital discharge
  New antibiotic therapy instituted after hospital discharge
30-day readmission rate | 30 days after hospital discharge
  Hospital readmissions up to 30 days after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Magnus N Lyngbakken, MD PhD, Principal Investigator — University Hospital, Akershus
Locations (12):
- Norway (12):
  - Haukeland University Hospital, Bergen
  - Drammen Hospital, Vestre Viken Hospital Trust, Drammen
  - Bærum Hospital, Vestre Viken Hospital Trust, Gjettum
  - Sykehuset Østfold HF, Grålum
  - Sørlandet sykehus HF, Kristiansand
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Ullevål, Oslo
  - Telemark Hospital Trust, Skien
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St. Olavs hospital, Trondheim
  - Sykehuset i Vestfold HF, Tønsberg

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-12-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT05045612/Prot_003.pdf
  • Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT05045612/SAP_001.pdf